CLINICAL TRIAL: NCT01939730
Title: Rituximab (IDEC-C2B8) Plus GM-CSF in Patients With Follicular B-Cell Lymphoma
Brief Title: Rituximab + GM-CSF in Patients With Follicular B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM98-304
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma
Keywords: Lymphoma; Follicular B-Cell Lymphoma; Rituximab; Rituxan; GM-CSF; Sargramostim; Leukine
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab + GM-CSF (Experimental): All patients receive one (1) course of therapy consisting of four (4) doses of rituximab, a single dose 375 mg/m^2 administered once weekly for 4 weeks along with GM-CSF 250 mcg subcutaneously three times weekly (tiw) for 8 weeks, starting 1 hour before the first dose of rituximab. In selected cases, the GM-CSF starts 1 week before, or 1 day after, the first rituximab dose.
  Interventions: Drug: Rituximab; Drug: GM-CSF

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2 by vein once a week for 4 weeks on Days 1, 8, 15, 22.
  Other Names: Rituxan
Drug: GM-CSF — 250 mcg subcutaneously 3 times a week for 8 weeks.
  Other Names: Sagramostim; Leukine

SUMMARY:
The goal of this clinical research study is to see if using the drugs Rituximab (IDEC-C2B8) and Granulocyte-macrophage colony-stimulating factor (GM-CSF) (Leukine) together is better than using rituximab alone to treat follicular B-cell lymphomas. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Rituximab seeks out and helps destroy cancer cells. GM-CSF stimulates the body to produce white blood cells.

Before treatment starts, patients will have a complete exam, including blood and urine tests. A chest x-ray and a CT scan or MRI scan of the abdomen and pelvis will be done to measure tumors. Bone marrow and lymph node samples will be taken.

Women who are able to have children must have a negative blood pregnancy test.

Patients in this study will receive both rituximab and GM-CSF. The combined treatment will last 8 weeks.

Rituximab will be given through a needle in a vein over 3-6 hours once a week. GM-CSF will be given through a needle under the skin 3 times a week. The first of these 3 doses will be usually given 1 hour before the rituximab dose. In selected cases, GM-CSF will start 1 week before or 1 day after the rituximab.

Patients may also receive the drugs acetaminophen (Tylenol) and diphenhydramine hydrochloride (Benadryl) 30-60 minutes before each dose of rituximab. This will be done to ease side effects. Patients may need to stay in the clinic for up to 2 hours after rituximab is given.

If the combined Rituximab and GM-CSF treatment causes severe side effects, the treatment may be stopped.

During the study, blood tests will be done before each rituximab treatment and after the first and fourth rituximab treatments. About 2 to 6 teaspoons of blood will be drawn for each test. A physical exam and a urine test will be done before the fourth rituximab treatment.

After all treatment is done, patients will have a complete exam, including blood tests once a week for 4 weeks and then at 2, 3, 6, 9, 12, 18, and 24 months. A CT scan or MRI scan of the abdomen and pelvis will also be done at 2, 3, 6, 9, 12, 18, and 24 months. Bone marrow samples will be taken at 2, 3, and 12 months. Some patients may also have bone marrow samples taken once a year after that. A large needle will be used to take the bone marrow samples.

This is an investigational study. GM-CSF and rituximab are approved for commercial use by FDA. As many as 40 patients will take part in the study. All will be treated as outpatients. The study will take place only at the University of Texas (UT) MD Anderson Cancer Center (MDACC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed follicular B-cell lymphoma. This can include relapsed patients, who have had no prior rituximab therapy, or previously untreated patients. Previously untreated patients should be made aware of higher priority protocols such as combination chemo-immunotherapy protocols, but if they decline that, they can be entered on this protocol.
2. Males or females, 18 years or older; expected survival of =/> 4 months; performance status of 0, 1 or 2.
3. Demonstrable monoclonal cluster of differentiation antigen 20 (CD20)-positive B-cell population.
4. Acceptable hematologic status including:

i. hemoglobin (Hgb) =/> 8.0 gm/dL

ii. White blood count (WBC) =/> 3.0 x 10^3/mm^3(x 10^9/L)

iii. Absolute granulocyte count =/> 1.5 x 10^3/mm^3

iv. Platelet count =/>75 x 10^3/mm^3

e. Adequate renal function (serum creatinine ≤ 2mg/dl)

Exclusion Criteria:

1. presence of Central Nervous System (CNS) Lymphoma
2. chronic lymphocytic leukemia (CLL)
3. small lymphocytic lymphoma
4. therapy in prior 3 weeks (6 weeks for nitrosourea; 6 months for Bone Marrow Transplantation (BMT))
5. patients who received prior rituximab or other anti-CD20 therapy
6. serious non-malignant disease, or other malignancy
7. active infection
8. history of HIV infection

i pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1999-08; Primary Completion 2006-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate of Rituximab plus GM-CSF of repeat doses (once weekly times four) | 1 month
  Response Rate is the number of participants with response compared to total. Response definitions: Complete response (CR) defined as those who achieve a normal state which includes no detectable evidence of disease on x-rays. Complete response "unconfirmed" (CRu) defined on the basis of minimal residual abnormalities on x-ray such as a residual mass <25% of original measurement with no palpable disease on physical examination. Partial response (PR) defined as 50-75% reduction in the product of palpable tumor diameters of in the tumor volume measurements by radiologic criteria or any palpable disease such as peripheral node(s) > 1 cm in diameter or palpable abdominal mass with histological evidence of lymphoma cells. Minor response or failure includes <50% tumor shrinkage, or > 50% but with tumor regrowth between courses.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Samaniego, MD, MPH, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org